CLINICAL TRIAL: NCT06857539
Title: The ELEVATE Program for Prediction, Early Detection & Intervention in Cerebral Palsy
Brief Title: Assessing Intellectual and Motor Outcomes in High-risk Infants
Acronym: AIM-High
Status: Not yet recruiting | Type: Observational
Sponsor: University College Cork (Other)
Collaborators: Coombe Women and Infants University Hospital (Other); The Rotunda Hospital (Other); Cerebral Palsy Foundation (Unknown); Karolinska Institutet (Other); University of Pisa (Other); Göteborg University (Other)
Responsible Party: Principal Investigator, Dr. Deirdre Murray, Professor of Paediatrics, University College Cork
Other Study IDs: DM01
Record Dates: First submitted 2024-12-05; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Palsy; Cerebral Palsy (CP); Cerebral Palsy Children; High-risk Infants; Intellectual and Developmental Disabilities; Motor Impairment; Cognitive Development
Keywords: Cerebral Palsy; High-Risk Infant Follow-up; Motor Difficulty; Intellectual Delay; Cognitive Impairment
MeSH Terms: conditions — Cerebral Palsy; Developmental Disabilities; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Months
Biospecimen Retention: Samples Without DNA — Microsampling will be used to collect samples from high-risk infants in the neonatal unit. These will be used for biomarker analysis including neurospecific proteins and mRNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- High-Risk Group: This group will have risk factors such as prematurity or hypoxic-ischaemic encephalopathy which put them in the High-Risk cohort
- Control Group: This group will be healthy, term infants who do not require admission to neonatal intensive care

SUMMARY:
Cerebral palsy (CP) is a condition when a baby has a brain injury that affects their movement and muscle tone. Some people with CP can have other developmental issues, like learning impairments, but many do not and have isolated issues with their motor skills. Some newborns are at higher risk of developing CP, including babies born prematurely, those who have an injury to their brain, and those who have an abnormal neurological examination. However, most babies with a higher risk of CP do not develop CP. The problem is that doctors can't tell early on who will and who will not develop CP, they can only say who has a risk of it. Therefore, these babies are followed up in out-patient clinics to see how they are progressing, usually by a neonatologist (baby doctor), often a physiotherapist, and some may also be referred to services in the community like the Early Intervention Team. If there is a significant concern, doctors will often perform a scan of the baby's brain to provide more information. Even with all this follow-up, it still usually takes at least 12 months, and can be up to 2 years, to diagnose a child as having CP.

In this study the aim is to try and reduce the age of diagnosis of CP by assessing children in high-risk out-patient clinics using novel and specific examinations. This study is being conducted at several hospitals in Ireland, including Cork University Maternity Hospital (CUMH), The Rotunda Hospital and the Coombe Women and Infants Hospital. It is being coordinated by the In4kids network and will be conducted in the INFANT Centre/ University College Cork (UCC). The study has been funded by Science Foundation Ireland (SFI) and the Cerebral Palsy Foundation, USA.

ELIGIBILITY:
Inclusion Criteria:

- (High Risk Group)

Legal guardians must be able and willing to give written informed consent and to comply with the requirements of this study protocol.

All infants considered high risk for a diagnosis of cerebral palsy and neuro-developmental impairment will be eligible, specifically including:

All preterm infants born ≤32 weeks Post Menstrual Age or ≤1500 gm birth weight

All encephalopathic infants

Neurological risk factors (e.g., cerebral birth defect, injury/malformation on neuroimaging, persistently abnormal neurological exam)

(Control Group)

All full term infants will be eligible if:

Term infants born > 37 weeks gestational age

Not admitted to the NICU

No neurological impairments at birth (no identified congenital or genetic abnormalities)

Exclusion Criteria:

- (High Risk & Control Groups)

Death prior to discharge from the neonatal unit (High-Risk Infants only)

No parental consent (High-Risk and Control Infants)

Ages: 0 Days to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All infants considered high risk for a diagnosis of cerebral palsy and neuro-developmental impairment will be eligible, specifically:
  All preterm infants born ≤32 weeks Post Menstrual Age or ≤1500 gm birth weight
  All encephalopathic infants
  Neurological risk factors (e.g., injury/malformation on neuroimaging, persistently abnormal neurological exam)
  All full-term infants (>37 weeks gestation), without requirement for admission to the NICU will be eligible to be enrolled in the study as the control arm of the study
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-03-04 (Estimated); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
A | From near term to 4 months corrected gestational age
  To characterise the development of neural architecture and function during sleep using EEG, from the near-term period to 4 months corrected gestational age for infants at elevated risk of cerebral palsy and diagnosed with cerebral palsy
B | Birth to 6 weeks
  To examine underlying neuro-specific protein profiles near term corrected gestational age as early biomarkers of altered neural function, motor and developmental outcomes in infants at elevated risk of cerebral palsy and diagnosed with cerebral palsy.
C | 4 to 24 months
  Develop novel measures of cognitive outcome, including executive function, and use these to compare trajectories in infants with cerebral palsy and those without, from 4 to 24 months

SECONDARY OUTCOMES:
A | During the study period, ie. over five years
  To optimise existing predictive machine learning algorithms
B | 4 months
  To develop and establish a standardised, early fixation classification assessment tool that can be used for infants at risk of cerebral palsy in high-risk follow-up clinics across Ireland
C | 18 months
  To investigate ophthalmological biomarkers, including morphology, as potential early predictors of cerebral palsy and cognitive outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre M Murray, Principal Investigator — INFANT Research Centre, University College Cork, Cork, Ireland
Locations (4):
- Ireland (4):
  - Cork University Maternity Hospital, Cork
  - INFANT Centre, University College Cork, Cork
  - Coombe Women and Infant's Hospital, Dublin
  - The Rotunda Hospital, Dublin

IPD SHARING:
Plan to Share IPD: No
Individual Patient Data may not be shared according to ethical approval

REFERENCES:
- See also: Launch of Cerebral Palsy Research Programme at University College Cork — https://www.infantcentre.ie/2024/03/22/tanaiste-launches-new-e11-6-million-cerebral-palsy-research-programme-at-university-college-cork/
- See also: Inaugural lecture: Professor Deirdre Murray, CPF Chair in Early Brain Injury and Cerebral Palsy — https://www.infantcentre.ie/2024/03/23/professor-deirdre-murray-inaugural-lecture/